CLINICAL TRIAL: NCT03399253
Title: A Prospective,Multicentral,Open-label,Randomized,Controlled,Phase III Clinical Trial of Chemotherapy Alone Versus D2 Gastrectomy and Metastasectomy Plus Chemotherapy for Distal Gastric Cancer With One Non-curable Factor
Brief Title: Chemotherapy Alone Versus Surgery Plus Chemotherapy for Distal Gastric Cancer With One Non-curable Factor
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCGC004
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Gastric Cancer
Keywords: Distal Gastric Cancer, Gastrectomy, Metastasectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Surgical Procedures, Operative; Drug Therapy; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy (Active Comparator): chemotherapy with capecitabine and oxaliplatin (eight 3-week cycles of oral capecitabine 1000 mg/m² twice daily on days 1-14 plus intravenous oxaliplatin 130 mg/m² on day 1) for 6 months or progress of disease
  Interventions: Drug: chemotherapy
- Surgery+Chemotherapy (Experimental): D2 Gastrectomy and Metastasectomy + chemotherapy with capecitabine and oxaliplatin (eight 3-week cycles of oral capecitabine 1000 mg/m² twice daily on days 1-14 plus intravenous oxaliplatin 130 mg/m² on day 1) for 6 months or progress of disease
  Interventions: Procedure: surgery; Drug: chemotherapy

INTERVENTIONS:
Procedure: surgery — D2 gastrectomy + metastasectomy
  Arms: Surgery+Chemotherapy
Drug: chemotherapy — capecitabine and oxaliplatin (eight 3-week cycles of oral capecitabine 1000 mg/m² twice daily on days 1-14 plus intravenous oxaliplatin 130 mg/m² on day 1) for 6 months or progress of disease
  Other Names: XELOX

SUMMARY:
Our study aims to compare the efficacy and safety of Chemotherapy Alone Versus D2 distal gastrectomy and metastasectomy plus Chemotherapy for gastric cancer (GC) with one non-curable Factor

DETAILED DESCRIPTION:
Gastric cancer is the fourth most common malignancy worldwide and the second leading cause of cancer-related deaths, with the highest mortality rates reported in East Asia, including China. Many patients are diagnosed at an advanced stage of gastric cancer because of late onset and nonspecific symptoms. The prognosis of patients with advanced gastric cancer with non-curable factors, such as hepatic, peritoneal, or distant lymph node metastases, is poor. Chemotherapy is the standard of care for these patients. Palliative resection or bypass surgery is generally indicated in the presence of major symptoms such as bleeding or obstruction for incurable advanced gastric cancer. The usefulness of gastrectomy and metastasectomy is still unclear.

The REGATTA trial is the first clinical trial to explore the significance of surgery for incurable advanced gastric cancer. However, it concluded an opposite conclusion that gastrectomy followed by chemotherapy did not show any survival benefit compared with chemotherapy alone in advanced gastric cancer with a single non-curable factor. Interestingly, there was a significant interaction between treatment effect and tumor location in subgroup analyses of overall survival. Gastrectomy plus chemotherapy was associated with significantly worse overall survival in patients with upper-third tumors for less chemotherapy cycles. This finding raises the question whether inclusion criteria were restricted to the patients with lower-third tumor, findings of study might have been positive. So we raise this new trail to assess the significance of Gastrectomy and Metastasectomy for Distal Gastric Cancer With One Non-curable Factor.

ELIGIBILITY:
Inclusion Criteria:

1. Lower age limit of research subjects 18 years old and upper age limit of 75 years old.
2. PS (ECOG) of 0 or 1.
3. Without any other malignancies.
4. Written informed consent from the patient.
5. Standard gastrectomy with D2 lymphadenectomy for primary cancer
6. A single non-curable factor was defined by preoperative CT :

   hepatic metastasis (H1 or H2; maximum diameter ≤4 cm, number ≤4); peritoneal metastasis (R0 or R1 resection) para-aortic lymph node metastasis （number ≤4) ovarian metastasis adrenal metastasis renal metastasis
7. No contraindications to chemotherapy, including normal peripheral blood routine, liver and kidney function and electrocardiogram （WBC≥4.0 x 109 /L, NEU≥1.5 x 109 /L,PLT≥100 x 109 /L and HGB≥90g/L)

Exclusion Criteria:

1. Female in pregnancy or lactation.
2. Supraclavicular lymph nodes metastases，lung and bone metastases.
3. Massive ascites or cachexia.
4. Extensive cancer metastases of liver, peritoneal metastasis,para-aortic lymph node
5. Patients participating in any other clinical trails currently，or participated in other trails within 1 months.
6. Suffering from other serious diseases, including cardiovascular, respiratory, kidney, or liver disease, complicated by poorly controlled hypertension, diabetes, mental disorders or diseases.
7. Poor treatment compliance of patients
8. The group of chemotherapy alone accepts gastrectomy for bleeding or obstruction
9. Failure of R0 or R1 metastasectomy and gastrectomy with D2 lymphadenectomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-12-10 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5-year
  OS

SECONDARY OUTCOMES:
progression free survival | 3-year
  PFS

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Xu, PHD, Principal Investigator — Sun Yat-sen University
Locations (9):
- China (9):
  - Anqing Municipal Hospital, Anqing, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Cancer Center of Sun Yat-sen University, Guangzhou, Guangdong
  - Yuebei People's Hospital, Guangzhou, Guangdong
  - Jiangxi Provincial Cancer Hospital, Nanchang, Jiangxi
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin